CLINICAL TRIAL: NCT07345286
Title: Aspects Cliniques, Prise en Charge et Surveillance Des Maladies fébriles en RDC
Brief Title: Clinical Aspects, Management and Surveillance of Febrile Illnesses in DRC
Acronym: FI-CARE
Status: Recruiting | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: 1822/24
Record Dates: First submitted 2025-05-09; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Febrile Illness Acute; Biomarkers; Surveillance
Keywords: febrile illness; CRP; biomarkers; surveillance; clinical characteristics; Subsaharan Africa; malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma full blood treated with DNA/RNA shield
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with febrile illness: Patients with febrile illness matching inclusion/exclusion criteria presenting at emergency department or outpatient clinic. At this moment one site has been selected. Other sites might be added in the future given rise to other cohorts of febrile patients

SUMMARY:
The epidemiology and outcome of febrile illnesses in the Democratic Republic of Congo (DRC) is poorly documented. The FIKI² study, a prospective observational study of community-acquired febrile illnesses coordinated by ITM and INRB and conducted at 2 clinical sites from 2021 to 2023, has deepened the knowledge of clinical presentation, etiology, outcome and profile of inflammatory/infectious biomarkers (white blood cells and C-reactive protein, or CRP).

The management of febrile illnesses remains fraught with clinical challenges. Overuse of antibiotics in primary care remains a reality in the field, and has been observed in several studies, including FIKI². A number of initiatives are underway to address this problem, such as the use of biomarkers, the development of treatment guidelines and electronic decision support systems. The FIKI² study highlighted the potential role of CRP in rationalizing antibiotic use. In parallel, the 'AWARE antibiotic book' was published at the end of 2022 by the WHO, providing recommendations on the choice (or otherwise) of antibiotic therapy for over 30 common clinical infections, in both primary care and hospital settings.

Based on the results of the FIKI² study, the main aim of the FI-CARE study is to investigate the impact of these new tools (CRP biomarker, AWARE antibiotic book, and electronic decision support systems) on first-line antibiotic use. Secondly, the study will consolidate previous results from FIKI² sites in terms of monitoring the etiologies of community-acquired febrile illnesses (particularly arboviruses); and reinforce this monitoring at new sites (depending on opportunities). This complementary study will also pursue FIKI²'s strategic objectives of strengthening clinical research capacity and consolidating biobanks in the DRC.

FI-CARE is a prospective, observational, multicenter cohort study of adults and children presenting to the emergency department or outpatient clinic with community-acquired febrile illness. A laboratory component with sample storage in a biobank is added in a modular fashion according to laboratory and research capacities, epidemiological interest and available funds.

DETAILED DESCRIPTION:
The management of febrile illnesses in low resource settings remains fraught with clinical challenges. Overuse of antibiotics in primary care remains a reality in the field, and has been observed in several studies. A number of initiatives are underway to address this problem, such as the use of biomarkers, the development of treatment guidelines and electronic decision support systems. The 'AWARE antibiotic book' was published at the end of 2022 by the WHO, providing recommendations on the choice (or otherwise) of antibiotic therapy for over 30 common clinical infections, in both primary care and hospital settings.

As in most sub-Saharan African countries, very little data is available in the Democratic Republic of Congo (DRC) on the epidemiology, clinical presentation, causes and outcome of febrile illnesses, and research capacity is generally very weak.

FIKI² was a bi-centric observational study of febrile illnesses conducted between March 29, 2021 and October 9, 2023 at two newly established research sites in the DRC: (i) the pediatric emergency department of the Hôpital Général de Référence de Kinshasa (HGRK) - now the Centre Hospitalier Universitaire Renaissance (CHUR) - , and (ii) the emergency and outpatient department of the Hôpital Général de Référence (HGR) of the Institut Médical Evangélique (IME) in Kimpese.

The study prospectively recruited patients presenting with fever and collected data on clinical and laboratory characteristics at the time of consultation and during a three-week follow-up period. The study included the routine performance of a thick smear and/or RDT for malaria, in line with routine care, as well as the performance of an RDT for dengue and the measurement of CRP, hemoglobin, white blood cell count and differentiation as study laboratory procedures.

The study was also integrated for part of its duration into a blood culture surveillance project (protocol approved in Belgium and DRC). Blood samples were also collected for long-term storage and secondary research during the second phase of the study for consenting patients.

The conduct of the study was integrated with research and clinical capacity building, focusing on clinical assessment and CRP evaluation in the management process, in order to reduce antibiotic overuse.

The study provided important insights into the clinical presentation of febrile illnesses, and confirmed the significant impact of malaria on CRP levels, as well as its discriminating value in cases of undifferentiated fever and non-malarial respiratory tract infection. It highlighted a relatively high frequency of fever-associated bacteremia in ambulatory patients (of unclear clinical significance). The study confirmed high rates of inappropriate antibiotic prescribing. While FIKI² was not an interventional study, it was observed that the implementation of CRP was progressively associated with a marked reduction in antibiotic use (especially in cases of undifferentiated fever and non-malarial respiratory tract infection with normal CRP levels), once this test was integrated into the reasoning of the investigating clinicians.

FI-CARE study is a new study that extends the FIKI² study in terms of consolidating epidemiological and etiological research, but has as new objectives to measure the impact of CRP and the AWaRe guide on clinical management (reduction in antibiotic prescribing) AND to integrate effective surveillance of febrile illnesses with epidemic potential into primary care. Similar data collection tools as the FIKI² study will allow comparative analyses between the 2 studies.

In the first instance, the study takes place at the known site of the pediatric emergency department of the 'Centre Hospitalier Universitaire Renaissance de Kinshasa' (CHUR, formerly HGRK). Other sites may be added in the future, depending on epidemiological interest, research capacity and available funding (compatible with the principle of FA5 funds as seed money that can be used to attract further funding). The study is conceptualized as a modular one, with different levels of research depending on the research capacity and level of funding available at the sites involved:

1. Descriptive clinical characterization, focusing on systematic evaluation of tools to improve management (syndromic approach with CRP, AWaRe antibiotic book, or new electronic support systems), and surveillance (relevance of clinical case definitions).
2. Analysis of inflammatory biomarkers: C-reactive protein (CRP), white blood cells and their differentiation using different types of point-of-care (POC) equipment: portable analyzers and RDTs.
3. Etiological investigation of specific febrile illnesses

   1. Blood culture surveillance: as part of a project to improve antibiotic resistance surveillance and clinical management (protocol approved in DRC and Belgium).
   2. Evaluation of arboviral pathogens using multiplex diagnostic tools: complementary to surveillance objectives. These analyses will be carried out on stored samples.
4. Storage of well-documented samples with clinical data, enabling subsequent development and evaluation of diagnostic and surveillance platforms, and other secondary post-hoc research. Future analyses may include transcriptional profiling of peripheral blood to search for early biomarkers to distinguish bacterial from viral infections.

Study procedures are as follows:

* prospective recruitment of patients presenting with fever
* data collection on clinical and laboratory characteristics at the time of consultation and during a three-week follow-up period
* blood sampling at inclusion for routine analyses, performance of a thick smear and/or RDT for malaria, in line with routine care, as well as measurement of CRP, hemoglobin, white blood cell count and differentiation as study laboratory procedures; and for sample storage
* biobanking of relevant samples (plasma and full blood treated with DNA/RNA shield) for arboviral multiplex PCR and secondary analyses

ELIGIBILITY:
Inclusion Criteria:

* Ongoing fever objectified at presentation, or documented at home or other health center within 24 hours prior to presentation, defined as: axillary or tympanic temperature > 37.5°C, or oral or rectal temperature > 38°C.
* Opportunity for contact between patient (or designated relative) and study team on days 7, 14 and 21.
* Informed consent to participate signed by the patient (adult) or a legally acceptable representative (child or patients whose condition does not allow them to sign informed consent), with the assent of children aged 12 and over, wherever possible.

Exclusion Criteria:

* Child less than two months old.
* Hospitalization of > 48h in the last 14 days.

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with febrile illness presenting at the study site
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Describe and compare the use of antibiotics for patients with community-acquired febrile illness with different types of support | at enrollment
  Describe and compare the use of antibiotics for patients with community-acquired febrile illness with different types of support that can be used throughout the study to guide patient management (e.g. algorithm combining presenting syndrome with CRP results; etiological approach based on the WHO clinical guide (AWARE antibiotic book) or other; or any new electronic decision-making support). Endpoints:
  Frequency of antibiotics and class of antibiotics used with different types of support
Describe the appropriateness of antibiotics for patients with community-acquired febrile illness with different types of support | at enrollment
  Describe the appropriateness of antibiotics for patients with community-acquired febrile illness with different types of support that can be used throughout the study to guide patient management (e.g. algorithm combining presenting syndrome with CRP results; etiological approach based on the WHO clinical guide (AWARE antibiotic book) or other; or any new electronic decision-making support). Endpoints:
  - Appropriateness of antibiotic use (according to local clinical guidelines if available or WHO)
Describe and compare adherence to different types of support used | at enrollment
  Describe and compare adherence to the tools used to guide patient management (syndromic algorithm; AWARE antibiotic book or other etiological guide; or an electronic decision support). Endpoints:
  - frequency of adherence to recommendations
Describe reasons for non-adherence to different types of support used | at enrollment
  Describe reasons for non-adherence to the tools used to guide patient management (syndromic algorithm; AWARE antibiotic book or other etiological guide; or an electronic decision support). Endpoints:
  - frequency of reasons for non-adherence
Describe clinical presentation of febrile illnesses in the DRC. | from enrollment to the end of the 3 week follow-up period
  endpoints:
  - Frequency of specific symptoms
Describe laboratory presentation of febrile illnesses in the DRC. | from enrollment to the end of the 3 week follow-up period
  endpoints:
  - Frequency of laboratory deviations
Describe severity of febrile illnesses in the DRC. | from enrollment to the end of the 3 week follow-up period
  endpoints:
  - frequency of presence of severity criteria
Describe etiology of febrile illnesses in the DRC. | from enrollment to the end of the 3 week follow-up period
  endpoints:
  - Frequency of specific and syndromic diagnoses
Evaluate the frequency of hospital admissions for febrile illnesses in the DRC. | from enrollment to the end of the 3 week follow-up period
  endpoints:
  - Proportion of patients with a primary or secondary hospital admission
Evaluate the frequency of secondary visits for febrile illnesses in the DRC. | from enrollment to the end of the 3 week follow-up period
  endpoints:
  - Proportion of patients with secondary visits
Describe outcome of febrile illnesses in the DRC. | from enrollment to the end of the 3 week follow-up period
  endpoints:
  - Proportion of participants resolved, unresolved and dead by day 21

SECONDARY OUTCOMES:
Describe the biomarker profile (CRP, white blood cell count with differentiation) at inclusion of patients with febrile illnesses, and its correlation with specific and syndromic diagnoses and outcome. | at inclusion
  endpoint: White blood cell and CRP levels at baseline overall and for different patient categories (specific diagnosis and outcomes)
Evaluate the field accuracy of clinical case definitions currently used for national surveillance of the epidemic-prone subgroup. | from enrollment to the end of the 3 week follow-up period
  Endpoint:
  proportion of cases meeting one of the case definitions for diseases under surveillance correlated with final diagnosis
Evaluate the timeliness of reporting for diseases under national surveillance, of the epidemic-prone subgroup. | from enrollment to the end of the 3 week follow-up period
  Endpoint:
  proportion of diseases under national surveillance, of the epidemic-prone subgroup reported to health authorities in time.

OTHER OUTCOMES:
Describe the frequency and etiology of community-acquired bacteremias detected in patients with febrile illness | at inclusion
  Endpoint:
  frequency of bacteremia and identified germs.
Describe the antibiotic resistance profiles of community-acquired bacteremias detected in patients with febrile illness | at inclusion
  Endpoint:
  frequency of antibiotic resistance profiles of identified germs causing bacteremia.
Describe the frequency of arboviral diseases detected by a specific PCR panel (initially Dengue, Chikungunya, Zika, Yellow Fever) | from enrollment to the end of the 3 week follow-up period
  Endpoint:
  - frequency of confirmed arbovirus pathogens
Describe clinical and biological presentation of arboviral diseases detected by a specific PCR panel (initially Dengue, Chikungunya, Zika, Yellow Fever) | from enrollment to the end of the 3 week follow-up period
  Endpoint:
  - frequency of specific clinical and laboratory predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bottieau, PhD, Principal Investigator — ITM
Locations (1):
- Centre Hospitalier Universitaire Renaissance, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
Anonymized study data will be supplemented by metadata and documentation, such as the study protocol, annotated CRFs and other information such as codes, which together constitute a dataset, but will not include any direct identifiers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study data relating to participants will be available for sharing within a reasonable time after the study and in accordance with ITM's research data sharing principles for a duration of 2O years.
Access Criteria: Researchers will be able to request access to anonymized data for well-defined research or secondary analysis via a controlled access procedure.
URL: https://www.itg.be/en/research/data-sharing-and-open-access